| Official Title: | An Assessment of TLR4 and TOPK/PRPK Signaling in Sun |
|---|---|
| | Damaged Human Skin Acutely Exposed to Solar Simulated |
| | Light |
| NCT number: | NCT05398237 |
| <b>Document Type:</b> | Consent Form |
| Date of the | Version 06/20/2022, IRB approved 7/12/2022 |
| Document: | |

#  Consent to Participate in Research

**Study Title:** An Assessment of TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin

Acutely Exposed to Solar Simulated Light

Principal Investigator: Clara Curiel, MD

**Sponsor:** National Institute of Health

**This is a consent form for research participation.** It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to participate.

# Why is this study being done?

The purpose of this project is to obtain clinical data, including skin samples, that will help investigators evaluate changes occurring in sun damaged human skin as a result of light that simulates sun exposure (Solar Simulated Light or SSL). Of specific interest are the molecular targets for cancer prevention. Molecular targets are the parts of the body's cells that have been shown to play a role in causing or preventing cancer and which scientists seek to affect in a way that may slow or eliminate the development of cancer.

# What will happen if I take part in this study?

First, you will be screened to see if you are eligible for the study. Screening includes discussing the study, reading and signing this Consent form, a skin exam, and a medical history review. Information collected during the phone-screening interview that was done when you first called the study coordinator will be used by the medical provider to determine if you are eligible for the study, and it may be used as study data for analysis.

If you are eligible to participate in the study, your first study Visit will be scheduled. In some cases, it may be possible to combine the screening visit and Visit 1 as a single appointment. Please see below for the schedule you will follow if you participate in this study:

#### Visit 1 – Will last about 1 hour

You will be assigned a study identification number, and the test areas on your left buttock will be outlined with non-permanent skin marking ink. If you are a woman of childbearing potential, a urine pregnancy test will be done at this visit. We will also determine the amount of solar simulated light (SSL) that will be used on your skin. This is called your Minimal Erythema Dose (MED). Since everyone responds differently to sunlight, we will expose 6 different doses of SSL on your left buttock. The solar simulator has a row of six openings, which can be carefully controlled to deliver different amounts of light to circles on the skin. Each opening is 3/8 inch in diameter. The six openings will be spaced in a row about 3½ inches in length in the test area. The exposure time will be one minute. Your next appointment will be scheduled to take place about 24 hours later.

| Subject Initials: | ID#: |
|-------------------|-----------------------------|
| | Consent Version: 06/20/2022 |

#### 

You will be given a study diary to write down any illness or injury you may have, any changes in medications or vitamin supplements, and your sun exposure during the study. A study coordinator will show you how to use the diary, which you will bring with you to each study visit.

# Visit 2 – Will last about 30 minutes and must occur 22 to 26 hours after Visit 1

Your MED test dose will be identified by selecting the lowest dose of SSL that produces even redness on the test circle at 22-24 hours after exposure.

## Visit 3 – Will last about 1.5 hours and may be combined with Visit 2 if possible

Three biopsy test areas will be marked on your left forearm with non-permanent surgical marking ink. One of the biopsy test areas will not be exposed to solar simulated light and will serve as the "control" sample. The other two test areas will be exposed to solar simulated light. The total exposure time will be 2 minutes.

The control biopsy test area and one of the SSL exposed test areas on your left forearm will be collected 1 hour after the SSL exposure. This procedure will be performed in the following manner: a small volume of local anesthetic (painkiller) will be injected into the skin at each test area to numb the area. A 3/8" diameter piece of skin will be removed and 2 or 3 stitches will be placed to close each site, which will be covered with a small bandage. You will need to keep the sites clean, dry and covered for 10-16 days. Prior to the biopsy, photographs of your left forearm will be taken and labeled with your study number, initials, and the date.

## Visit 4 – will last about 1 hour and must occur 22 to 26 hours after Visit 3

During this visit the third biopsy test area on your left forearm will be collected, using the same procedure as described above. Prior to the biopsy, photographs of your left forearm will be taken and labeled with your study number, initials, and the date. Your study diary will be reviewed.

#### Visit 5 – will last about 20 minutes and must occur 10 to 16 days after Visit 4

The stitches will be removed from all of the biopsy sites. If you prefer, you may also have your sutures removed by an outside provider. The study coordinator will also review your study diary with you and discuss any health concerns or medication changes that you may have experienced during the study.

#### How long will I be in this study?

Participation in the study involves 5 visits to the clinic over the course of 4 weeks.

#### How many people will take part in this study?

Up to 36 patients will be enrolled in this study.

# What risks, side effects, or discomforts can I expect from being in the study?

Since this study is designed to simulate sun exposure to small areas of skin, mild to moderate sunburn and tanned spots at the site of the simulated sunlight exposure is a risk. These areas, where not removed by biopsy, will fade over time. Brief discomfort may be felt when the local

| Subject Initials: | ID#: |
|-------------------|-----------------------------|
| | Consent Version: 06/20/2022 |

#### 

painkiller (lidocaine) is injected prior to skin biopsies; however, it is usually minimal. Some people experience discomfort from the biopsies despite the use of the painkiller, and there is a slight risk of an allergic reaction to the painkiller. There is a slight chance of infection following the biopsies. It is expected that you will have a small (1/4 - 1/2 inch) scar at the biopsy site(s), which may be permanent or may fade over time. In addition, rare complications associated with skin biopsies include moderate temporary bleeding, as well as a numbing sensation of the skin around the biopsy sites, which might or might not be reversible.

If unanticipated side effects happen during this study or any information becomes available that may affect your willingness to participate, you will be informed.

# What benefits can I expect from being in this study?

There is no direct benefit to you by being in this study. We hope the information learned from this study will benefit patients with cancer in the future.

# What happens if I am injured because I took part in this study?

Side effects (injury) can happen in any research study. These effects may not be your fault or the fault of the researcher involved. Known side effects have been described in the "What risks, side effects, or discomforts can I expect from being in the study?" section of this consent form. However, side effects that are not currently known may happen and require care.

If you experience an injury or unanticipated adverse event, please call Doctor Curiel at (520) 626-6024 immediately. You can request medical treatment if you are injured as a result of taking part in this study. You and/or your health plan will be charged for this treatment. This, however, does not waive your rights in the event of negligence. If you suffer an injury from participating in this study, you should seek treatment. The University of Arizona has no funds set aside for the payment of treatment expenses for this study.

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study. You do not give up any of your legal rights by signing this form.

# Can I stop being in this study?

**Your participation is voluntary.** If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with the University of Arizona. If you are a student or employee at the University of Arizona, your decision will not affect your grades or employment status.

# What other choices do I have if I do not take part in this study?

You can choose not to participate in this study. You will not experience penalty or loss of benefits to which you are otherwise entitled.

When may participation in the study be stopped?

| Subject Initials: | ID#: |
|-------------------|-----------------------------|
| | Consent Version: 06/20/2022 |

#### 

The medical provider may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- If you do not follow the study rules
- If the study is stopped by the sponsor, IRB, or FDA.

# What are the costs of taking part in this study?

There is no cost to you for being in this study other than your time.

You may be responsible for payment of any bills that your insurance may refuse to pay due to your participation in this research study.

# Will I be paid for taking part in this study?

You will receive \$275 at the end of the study, upon completion of all the required visits and tests. The amount of compensation will be prorated if you participate in the study for a shorter period of time. The prorated amount will be based upon the number of visits you complete out of a total of 5 visits. The visits that include biopsies will be compensated at a higher rate than visits that only involve SSL exposure or the removal of stitches. Specifically, you will receive \$40 for Visit 1, \$25 for Visit 2, \$110 for Visit 3, \$70 for Visit 4, and \$30 for Visit 5. There is no compensation for eligibility screening.

By law, payments to subjects may be considered taxable income. We are required to obtain your name, address, and Social Security number for federal tax reporting purposes. If your compensation for this research study or a combination of research studies is \$600 or more in a calendar year (January to December), you will receive an IRS Form 1099 to report on your taxes.

# Will my study-related information be shared, disclosed, and kept confidential?

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

| Subject Initials: | ID#: |
|-------------------|-----------------------------|
| | Consent Version: 06/20/2022 |

#### 

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

It is anticipated that there will be circumstances where your study-related information and protected health information (PHI) will be released to persons and organizations described in this form. If you sign this form, you give permission to the research team to use and/or disclose your PHI for this study. Your information may be shared or disclosed with others to conduct the study, for regulatory purposes, and to help ensure that the study has been done correctly. These other groups include:

- Office for Human Research Protections or other federal, state, or international regulatory agencies
- Food and Drug Administration (FDA)
- The University of Arizona (UA) and the UA Institutional Review Board, their agents or study monitors

Your PHI may no longer be protected under the HIPAA privacy rule once it is disclosed by the research team.

What study-related information and PHI will be obtained, used, or disclosed? Information related to this research study that identifies you and your PHI will be collected directly from you, and is considered "self-reported".

The PHI you are authorizing to be used and/or disclosed in connection with this research study:

- Name
- Address
- Contact details
- Date of birth
- Medical records
- Past medical history
- Family history
- Race
- Ethnic origin

Demographic information to be disclosed may include, but is not limited to, your name, address, phone number, or social security number. If you receive compensation for participating in this research study, information identifying you may be used or disclosed as necessary to provide that compensation. Your self-reported health records may include information related to the diagnosis or treatment of sexually transmitted diseases (STDs), acquired immunodeficiency syndrome (AIDS), human immunodeficiency virus (HIV), other communicable diseases, genetic information (e.g., genetic testing), and/or alcohol and/or drug abuse. The study staff and study sponsor's monitor may see this information while reviewing

| Subject Initials: | ID#: |
|-------------------|-----------------------------|
| | Consent Version: 06/20/2022 |

#### 

your regular health records for this study, but they WILL NOT create, collect, or disclose this type of information for the purposes of this research study.

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. Be aware that this Federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

# When will my authorization expire?

There is no expiration date or event for your authorization. Therefore, unless you cancel this authorization (as instructed below) this authorization will continue to be effective.

# Do I have to sign this authorization form?

You do not have to sign this authorization. However, if you decide not to sign, you will not be able to participate in this research study; and it will not affect any non-study medical treatment or health care, payment, enrollment in any health plans, or benefits.

# What do I need to know if I decide to cancel my authorization?

After signing the authorization, you may decide to cancel your previous authorization for the research team to use your PHI. If you cancel the authorization, you will no longer be able to stay in the research study. Please note that any PHI collected before you cancel the authorization may still be used. You may revoke the authorization by contacting the Principal Investigator in writing. Contact information is under "Who can answer my questions about the study?" at the end of this document.

#### Will access be limited to your research study record during this study?

You may not have access to the research information developed as part of this study until it is completed.

# Who can answer my questions about this study?

If at any time you feel you have had a research-related injury, or for questions, concerns, or complaints about the study you may contact Clara Curiel, MD, at (520) 694-6024.

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact Human Subjects Protection Program Director at 520-626-8630 or online at https://research.arizona.edu/compliance/human-subjects-protection-program.

If you are injured as a result of participating in this study or for questions about a study-related injury, you may contact Clara Curiel, MD, at (520) 694-6024.

To cancel your authorization for access to PHI you must notify the Principal Investigator in writing at the following address:

Clara Curiel, MD

| Subject Initials: | ID#: |
|-------------------|-----------------------------|
| | Consent Version: 06/20/2022 |


University of Arizona Cancer Center 3838 N. Campbell Ave. Tucson, AZ 85719

An Institutional Review Board responsible for human subjects research at The University of Arizona reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of participants in research.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Will my data or specimens be stored for future research?

**Specimens:** There may be some specimens (skin biopsy tissue) remaining after the study is complete. We would like to keep any of the specimens that are left over after the study for future research. These specimens will be stored in a central facility (called a "tissue bank") which is located here at the University of Arizona Cancer Center. Your sample will be stored there permanently and will not be available for use in making health care decisions for you. At some time in the future, your stored specimens may be used by other researchers for other tests that are not known at this time, including genetic research tests. Future research may include studies to learn more about skin cancer and its prevention. In most cases, you will not be told what your sample is being used for. You will not be contacted to provide additional information, and you will not be asked to provide samples in addition to those agreed upon in this consent form.

When your specimen(s) are sent to the researchers, samples will be identified by a unique study code. Researchers to whom the University of Arizona sends your sample and information will not know who you are. They must also sign an agreement that they will not try to find out who you are. If research results are published, your name and identifiable information will not be used.

If you are willing to allow the remaining specimens to be used for future research studies, you must specify your consent below. Consent for future use of your remaining samples is entirely voluntary and may be withdrawn at any time.

If you decide now that your specimens can be kept for research, you can change your mind at any time. Contact the Principal Investigator, Clara Curiel, M.D. at (520) 626-6024 and let her know that you do not want us to use your tissue, and it will no longer be used for research. If your specimen has already been used for research, it will not be possible to get it back.

Please read each sentence below and think about your choice. After reading each sentence, mark an X in the box for "Yes" or "No" and initial your choice. No matter what you decide to do, it will not affect your care.

| Subject Initials: | ID#: |
|---|---|
| My remaining specimens may be used in future research: Yes | |
| <b>Data:</b> The Skin Cancer Prevention Project at the University of Arizona a database of individuals who have been screened for a study by coresearch clinic. The purpose of the database is to be able to contact expressed an interest in participating in future studies. The data information and the information you provided to us when you were seen that the studies is to be able to contact expressed an interest in participating in future studies. | alling us or coming to the people who have already abase will include contact |
| You do not have to agree to become part of this database for fut participation in this study. If you do not give your consent, your inform of the database for participation in future studies. If you do condatabase, your information will still remain confidential to the externot be identified by name when the results of this study are published | mation will not become part assent to be included in the art required by law. You will |
| You may call the Study Coordinator at (520) 321-7747, if you have database and how it will be used. If you change your mind about bein you may contact the Principal Investigator, Clara Curiel, M.D. at (1) remove your name and records from the database for participation in | ng included in the database, 520) 626-6024 and we will |
| By marking the blank next to the "Yes" or "No" on the line below, blank, you are indicating your preference. | , and initialing the "initials" |
| ☐ Yes, include me in the database for future studies. Init | tials |
| $\square$ No, do not include me in the database for future studies. | tials |
| Signing the consent form I have read (or someone has read to me) this form, and I am aware the participate in a research study. I have had the opportunity to ask quest answered to my satisfaction. I voluntarily agree to participate in this is use and/or disclosure of my PHI. I am not giving up any legal rights by given a signed copy of this form. | stions and have had them study and I authorize the |
| Printed name of subject Signature of subject | Date |
| Investigator/Research Staff I have explained the research to the participant or the participant's rerequesting the signature(s) above. There are no blanks in this docume form has been given to the participant or to the participant's representation. | ent. A signed copy of this |
| Printed name of person Signature of person obtaining cor | nsent Date |

| Subject Initials: | ID#: |
|-------------------|-----------------------------|
| | Consent Version: 06/20/2022 |

obtaining consent